CLINICAL TRIAL: NCT06082752
Title: The Analysis of the Impact of 5-minute Massage Session on the Muscle Stiffness and Tone: a Randomised Control Trial
Brief Title: The Analysis of the Impact of 5-minute Massage Session on the Muscle Stiffness and Tone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Principal Investigator, Krzysztof Kassolik, Phd, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WroclawUHSS
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Musculoskeletal Disorder
Keywords: Massage therapy; Muscle tone; Muscle stiffness
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Experimental): In the intervention group measures will be taken twice: before and after the 5-minute massage session.
  Interventions: Procedure: Massage session
- Non-massage group (No Intervention): In the control group measures will be taken twice: at the beginning of the meeting and again after 5 minutes.

INTERVENTIONS:
Procedure: Massage session — Participants in the intervention group are provided with the 5-minute massage session in the medial and lateral gastrocnemius muscle (dominant leg).
  Arms: Massage group

SUMMARY:
The study design was a randomised, controlled, parallel, two-arm trial. The subjects were randomly assigned to one of the study groups: the intervention group or the control group. The passive mechanical properties, i.e. the stiffness and tone of the medial and lateral gastrocnemius muscle (dominant leg) were assessed. Measures were taken twice: in the intervention group before and after the 5-minute massage session, and in the control group at the beginning of the meeting and again after 5 minutes.

DETAILED DESCRIPTION:
The purpose of this study was to determine whether a 5-minute massage, applied to healthy individuals, may change the passive mechanical muscle properties, which supposedly may prevent MSDs. The study is carried out on the medial and lateral gastrocnemius muscles because of their accessibility and crucial role in locomotion. MyotonPRO and TMG S2 devices were used to assess the stiffness and radial muscle displacement of the gastrocnemius muscle respectively.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 24 years;
* healthy individuals, with no lower limb pathology;
* PA≥600 MET-min/week assessed by IPAQ questionnaire;
* no medical contraindication of massage therapy;
* body mass index 18,5 < BMI ≤ 25kg/m2
* signing the informed consent.

Exclusion Criteria:

* pregnant women;
* individuals suffering from neurologic or orthopaedic problems;
* lower limb surgical interventions;
* cancers;
* musculoskeletal disorders
* body mass index 18,5 > BMI ≥ 25kg/m2
* the lack of informed consent.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Changes in maximal displacement of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  The maximal radial displacement is produced in the muscle belly after the electrical stimulation. Measuring device: TMG S2
Changes in delay time of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  Delay time is the time in which the muscle displacement increases to 10% after the electrical stimulation. Measuring device: TMG S2
Changes in contraction time of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  Contraction time is the time between 10% and 90% of the muscle displacement after the electrical stimulation. Measuring device: TMG S2
Changes in sustain time of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  Sustain time is the time between 50% of maximum contraction to 50% of maximum relaxation of a muscle after the electrical stimulation. Measuring device: TMG S2
Changes in relaxation time of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  Relaxation time is the time between 90% of maximum contraction and 50% of maximum relaxation of a muscle after the electrical stimulation. Measuring device: TMG S2
Changes in oscillation frequency of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  The oscillation frequency characterizes the tension of muscle tissue. Measuring device: MyotonPRO
Changes in dynamic stiffness of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  The dynamic stiffness corresponds to the soft tissues' capacity to resist external forces. Measuring device: MyotonPRO
Changes in logarithmic decrement of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  Logarithmic decrement is the dissipation of the tissue oscillation. Measuring device: MyotonPRO
Changes in mechanical stress relaxation time of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  Mechanical stress relaxation time is the time needed for the muscle to recover to its initial shape. Measuring device: MyotonPRO
Changes in creep of the medial and lateral gastrocnemius muscle | 1) baseline, 2) immediately after the massage session
  Creep is the ratio of relaxation (R) and time between the beginning of the mechanical impulse and the time point of maximal displacement Measuring device: MyotonPRO

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Kassolik, Study Chair — Wroclaw University of Health and Sport Sciences
Locations (1):
- Wroclaw University of Health and Sport Sciences, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No